CLINICAL TRIAL: NCT06127615
Title: The Efficacy of the Longeviti ClearFit Implant in Craniectomies for Post-Operative Monitoring in Chronic Subdural Hematomas
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study did not enroll participants
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UKansasClearFit
Record Dates: First submitted 2023-10-03; First posted 2023-11-13 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-03

CONDITIONS: Chronic Subdural Hematoma
MeSH Terms: conditions — Hematoma, Subdural, Chronic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- ClearFit Longeviti Implant (Experimental): Patients with chronic subdural hematomas that qualify for study and agree to participate will receive the ClearFit implant to cover the craniectomy site and have ultrasound imaging for their post-operative follow-up rather than CT/MRI, with exception of first initial post-op CT scan, and crossover to CT/MRI if clinically indicated or required for diagnostic purposes/patient safety
  Interventions: Device: ClearFit

INTERVENTIONS:
Device: ClearFit — Implantation of ClearFit Longeviti Craniectomy Cover

SUMMARY:
Chronic subdural hematomas are frequent neurosurgical issues that are most often treated with burr hole craniectomies to drain the subdural fluid. At the chronic stage, a subdural hematoma is more liquified and easily washed out through burr hole openings. However, it often requires frequent imaging and monitoring to ensure that fluid does not reaccumulate in the subdural space, that the washout was adequate, and that further intervention/repeat intervention is not required, particularly if the patient develops acute changes in neurologic status or lacks improvement in initial symptomatology. Therefore, these patients require multiple repeated CT head images during their inpatient and post-operative follow-up course. This leads to high radiation doses to patients and high-cost burden. The Longeviti ClearFit Cover was developed to allow for ultrasound imaging through the implanted cover. The skull's acoustic properties prevent ultrasound from being used through the bone, therefore limiting its use in post-operative neurosurgical patients. Using ultrasound would remove the need for high radiation doses with CT, could be done very quickly and easily at bedside or in the clinic to check subdural space or ventricle size, and is much lower cost. This ClearFit implant would be utilized in place of a burr hole cover, typically titanium, that is implanted in most other cases. The aim of this study is to prospectively assess patients with surgically treated chronic subdural hematomas via craniectomy that have the craniectomy site covered with the Longeviti ClearFit, compared retrospectively to a matched cohort of patients that had their craniectomy site for the same procedure covered with the typically used titanium/metal. This will allow us to determine if this new implant results in reduced need for repeated CT imaging by utilizing bedside clinician-performed ultrasound and reduces overall cost for patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients >18 years old; patients determined by surgeon to have a chronic subdural hematoma that is treated with craniectomy that would allow for implantation of a ClearFit cover

Exclusion Criteria:

* Pediatric patients, patient with allergy to the material the implant is made with (polymethylmethacrylate)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Patient Radiation | from time of implant to last follow-up, anticipate 1 year
  Amount of radiation exposure to patient with ClearFit obtaining ultrasounds rather than CT compared to retrospective control group
Patient cost | from time of implant to last follow-up, anticipate 1 year
  Overall cost to patient with ClearFit compared to retrospective control group

SECONDARY OUTCOMES:
Quality of imaging | from time of implant to last follow-up, anticipate 1 year
  Calculated based on number of cross-overs from ultrasound to CT or MRI, with noted reason for crossover. Analysis of how often ultrasound is unable to be used/not feasible for post-operative monitoring of subdural, statistical analysis of crossover out of ultrasound into CT/MRI cranial imaging
Provider experience caring for patient | from time of implant to last follow-up, anticipate 1 year
  Survey of ease to care for patient in post-operative time period, ultrasound for imaging, transport of patient to obtain imaging, ease of access

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Belzberg M, Shalom NB, Yuhanna E, Manbachi A, Tekes A, Huang J, Brem H, Gordon CR. Sonolucent Cranial Implants: Cadaveric Study and Clinical Findings Supporting Diagnostic and Therapeutic Transcranioplasty Ultrasound. J Craniofac Surg. 2019 Jul;30(5):1456-1461. doi: 10.1097/SCS.0000000000005454. PMID 31299743
- [Background] Belzberg M, Shalom NB, Lu A, Yuhanna E, Manbachi A, Tekes A, Huang J, Brem H, Gordon C. Transcranioplasty Ultrasound Through a Sonolucent Cranial Implant Made of Polymethyl Methacrylate: Phantom Study Comparing Ultrasound, Computed Tomography, and Magnetic Resonance Imaging. J Craniofac Surg. 2019 Oct;30(7):e626-e629. doi: 10.1097/SCS.0000000000005651. PMID 31188246
- [Background] Hadley C, North R, Srinivasan V, Kan P, Burkhardt JK. Elective Sonolucent Cranioplasty for Real-Time Ultrasound Monitoring of Flow and Patency of an Extra- to Intracranial Bypass. J Craniofac Surg. 2020 May/Jun;31(3):622-624. doi: 10.1097/SCS.0000000000006225. PMID 32149973
- [Background] Flores AR, Srinivasan VM, Seeley J, Huggins C, Kan P, Burkhardt JK. Safety, Feasibility, and Patient-Rated Outcome of Sonolucent Cranioplasty in Extracranial-Intracranial Bypass Surgery to Allow for Transcranioplasty Ultrasound Assessment. World Neurosurg. 2020 Dec;144:e277-e284. doi: 10.1016/j.wneu.2020.08.114. Epub 2020 Aug 20. PMID 32827747
- [Background] Lee RP, Meggyesy M, Ahn J, Ritter C, Suk I, Machnitz AJ, Huang J, Gordon C, Brem H, Luciano M. First Experience With Postoperative Transcranial Ultrasound Through Sonolucent Burr Hole Covers in Adult Hydrocephalus Patients. Neurosurgery. 2023 Feb 1;92(2):382-390. doi: 10.1227/neu.0000000000002221. Epub 2022 Nov 15. PMID 36637272
- [Background] Doron O, D'Amico RS, Langer DJ. The Cranial Window: Opportunities for the Use of Bedside Ultrasound Facilitated by Sonolucent Implants in Neurosurgical Patients. World Neurosurg. 2022 Sep;165:142-144. doi: 10.1016/j.wneu.2022.05.084. Epub 2022 May 23. No abstract available. PMID 35926403
- [Background] Niesen WD, Rosenkranz M, Weiller C. Bedsided Transcranial Sonographic Monitoring for Expansion and Progression of Subdural Hematoma Compared to Computed Tomography. Front Neurol. 2018 May 28;9:374. doi: 10.3389/fneur.2018.00374. eCollection 2018. PMID 29892260
- See also: Related Info — https://www.sealedenvelope.com/power/binary-noninferior/